CLINICAL TRIAL: NCT01047527
Title: An Effectiveness Trial of Maintenance Therapy for Nicotine Dependence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Robert Schnoll, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DESPR DA025078; R01DA025078-02 (NIH)
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Results first posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-06

CONDITIONS: Nicotine Dependence
Keywords: nicotine replacement therapy, smoking cessation, transdermal nicotine
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 8 weeks transdermal nicotine (Active Comparator): 8 weeks of transdermal nicotine
  Interventions: Drug: Transdermal nicotine patch
- 24 weeks transdermal nicotine (Active Comparator): 24 weeks of transdermal nicotine
  Interventions: Drug: Transdermal nicotine patch
- 52 weeks transdermal nicotine (Experimental): 52 weeks of transdermal nicotine
  Interventions: Drug: Transdermal nicotine patch

INTERVENTIONS:
Drug: Transdermal nicotine patch — Transdermal nicotine, 21mg/day

SUMMARY:
The transdermal nicotine patch is the most widely used form of tobacco dependence treatment in the US and Europe, but most smokers are unable to successfully quit with this form of treatment. Failure to respond to this treatment may, to a large extent, be due to the use of nicotine patches for only 8 weeks, the recommended treatment duration. We have found in a controlled randomized clinical trial that using the nicotine patch for 24 weeks can increase quit rates significantly. We propose here a clinical trial to replicate and extend these results to a community setting in the real-world, using the same research design utilized in clinical trials to demonstrate the effectiveness of methadone maintenance therapy for opiate dependence. Specifically, 540 smokers will receive counseling and standard (8-weeks), extended (24-weeks), or maintenance (52 weeks) therapy with transdermal nicotine patches. The main outcome is biochemically-verified smoking cessation at week 52. The cost-effectiveness, safety, and mechanism of effect (e.g., promotion of recovery following a lapse) for maintenance therapy with transdermal nicotine will also be assessed. The study results may change how we treat nicotine dependence with transdermal nicotine.

DETAILED DESCRIPTION:
The transdermal nicotine patch is the most widely used form of tobacco dependence treatment in the US and Europe. Yet, abstinence rates following patch treatment are only ~20% at 6-months and ~9% at 12-months. There is a growing recognition that nicotine dependence is a chronic disease, like asthma or diabetes, which requires maintenance therapy. While current guidelines established by the USDHHS's Public Health Service (PHS) recommend 8-week duration for transdermal nicotine therapy, support for this recommendation is limited. In a recent randomized placebo-controlled efficacy trial comparing standard (8-week) vs. extended (24-weeks) treatment with nicotine patches, we found that, at 24 weeks, point-prevalence abstinence rates were 30% in the 24-week arm vs. 20% in the standard therapy arm (p < .05); however, by week 52, 6 months after treatment was discontinued for the extended treatment arm, the quit rates were equivalent across the treatment arms. This was the first clinical trial to suggest that the benefits of extended treatment with transdermal nicotine are largely dependent on the continuation of active treatment. However, as an efficacy trial, this study was conducted under highly-controlled conditions with strict inclusion/exclusion criteria to enhance internal validity. If recommendations for the duration of nicotine patch therapy are to be formally revised to encourage maintenance therapy, these findings must be replicated and extended under "real-world circumstances" in an effectiveness trial. In addition, as done in clinical trials to support the use of methadone maintenance for opiate dependence, a replication study must include a treatment arm that receives maintenance therapy throughout the duration of the trial (52 weeks). Thus, we propose to conduct a randomized effectiveness trial to evaluate the benefits of maintenance therapy with transdermal nicotine patches for smoking cessation. Specifically, 540 smokers will receive brief counseling and will be randomized to: standard (8-weeks), extended (24-weeks), or maintenance (52 weeks) transdermal nicotine therapy. The primary outcome will be biochemically verified 7-day point prevalence abstinence at week 52. Additional study aims include assessing: 1) treatment side effects across study arms; 2) longitudinal patterns of relapse and recovery across treatment arms; 3) mediators and moderators of treatment effects; and 4) cost-effectiveness. Overall, the trial findings will provide critical data for future PHS reviews of maintenance therapy with transdermal nicotine for subsequent treatment guidelines; for third-party payer assessments of maintenance transdermal nicotine as a covered benefit; and for individual smokers' decisions to use maintenance transdermal nicotine through over-the-counter access. In turn, this study may help to attain the Healthy People 2010 goals of reducing the US rate of tobacco use.

ELIGIBILITY:
Inclusion Criteria: Participants will be: 1) males and females over age 18 who smoke at least 10 cigarettes/day; 2) able to communicate in English; 3) able to use NRT safely (e.g., no allergy to latex, no serious abnormal ECG reading); 4) able to provide written informed consent for study procedures; and 5) residing in the geographic area for at least 12 months.

Exclusion Criteria: Participants will be ineligible for the trial if they: 1) are unable to communicate in English; 2) Have a current diagnosis of psychosis and/or manic depression; 3) have a current medical condition that would make using transdermal nicotine patch unsafe (e.g., allergy to latex, serious, abnormal ECG reading)- participants with asthma, diabetes, hypertension, or heart disease (e.g., coronary artery disease, abnormal heart rhythm, an arrhythmia) will be permitted to enroll in the study with medical clearance from the participant's physician or the study physician; 4) have had a heart attack within the past 6 months, 5) are pregnant or planning to become pregnant or lactating, or 6) are currently enrolled or plan to enroll in another research or smoking cessation program within the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2009-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Hitsman, PhD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Theodoulou A, Chepkin SC, Ye W, Fanshawe TR, Bullen C, Hartmann-Boyce J, Livingstone-Banks J, Hajizadeh A, Lindson N. Different doses, durations and modes of delivery of nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2023 Jun 19;6(6):CD013308. doi: 10.1002/14651858.CD013308.pub2. PMID 37335995
- [Derived] Schnoll RA, Goelz PM, Veluz-Wilkins A, Blazekovic S, Powers L, Leone FT, Gariti P, Wileyto EP, Hitsman B. Long-term nicotine replacement therapy: a randomized clinical trial. JAMA Intern Med. 2015 Apr;175(4):504-11. doi: 10.1001/jamainternmed.2014.8313. PMID 25705872

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 8 Weeks Transdermal Nicotine | 24 Weeks Transdermal Nicotine | 52 Weeks Transdermal Nicotine
Started | 180 | 173 | 172
8 Weeks | 148 | 142 | 138
24 Weeks | 111 | 123 | 119
Completed | 95 | 112 | 107
Not Completed | 85 | 61 | 65

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 8 Weeks Transdermal Nicotine | 24 Weeks Transdermal Nicotine | 52 Weeks Transdermal Nicotine | Total
Number analyzed (Participants) | 180 | 173 | 172 | 525
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (12.3) | 46.9 (12.2) | 46.4 (12.1) | 46.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 95 | 81 | 266
  Male | 90 | 78 | 91 | 259

OUTCOME MEASURES:

1. Primary Outcome: Point Prevalence Abstinence
Description: self-reported abstinence from smoking for 7 days prior to the assessment and biochemically confirmed with breath carbon monoxide
Time Frame: 52-week
Population: The primary objective of this study was to examine the benefits in terms of cessation of 52-weeks of treatment compared to 8 or 24 weeks.
Measure: Number; unit: participants
Groups:
- Standard + Extended: participants on standard or extended therapy
- Maintenance: Participants on 52 weeks of therapy
Arm/Group | Standard + Extended | Maintenance
Number analyzed (Participants) | 353 | 172
participants | 84 | 35

2. Primary Outcome: Week 24 Point Prevalence Abstinence
Description: as for outcome 1
Time Frame: 24-week
Population: This analysis was planned to replicate the previous study (Schnoll et al., 2010; Annals of Internal Medicine).
Measure: Number; unit: participants
Arm/Group | Standard | Extended + Maintenance
Number analyzed (Participants) | 180 | 345
participants | 39 | 94

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | 8 Weeks Transdermal Nicotine | 24 Weeks Transdermal Nicotine | 52 Weeks Transdermal Nicotine
Serious Adverse Events (participants affected / at risk) | 4/180 | 2/173 | 8/172
Other Adverse Events (participants affected / at risk) | 0/180 | 0/173 | 0/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8 Weeks Transdermal Nicotine (N=180) | 24 Weeks Transdermal Nicotine (N=173) | 52 Weeks Transdermal Nicotine (N=172)
Leg infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ovarian cysts (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Ductal Carcinoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Kidney Disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
High Blood pressure/cholesterol/blood clots (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
COPD/Pneumonia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Kidney Stones (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Calculus of Galbladder; chlecystits; pneumonia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Severe Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Lack of placebo; low adherence to nicotine patches; nicotine patches are not the most effective treatment for nicotine dependence; participant attrition was high.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes